CLINICAL TRIAL: NCT05028829
Title: Multi-center Double Blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of Long-term Atorvastatin (20 mg/Day) v. Placebo on HCC Risk in Individuals With Advanced Liver Fibrosis
Brief Title: Safety and Efficacy of Atorvastatin v. Placebo on HCC Risk
Acronym: TORCH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Raymond Chung (Other)
Collaborators: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor-Investigator, Raymond Chung, Director of Hepatology, MGH, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 21-444
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Liver Fibroses; Cirrhosis
Keywords: Liver Disease; Chemoprevention; HCC; Atorvastatin
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis; Liver Diseases | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Atorvastatin 20 mg (Experimental): Atorvastatin 20mg will be administered daily via oral route for 48 consecutive weeks on an outpatient basis.
  Interventions: Drug: Atorvastatin 20mg
- Group B: Placebo to Match (PTM) (Placebo Comparator): PTM will be administered daily via oral route for 48 consecutive weeks on an outpatient basis.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin 20mg — Oral administration of atorvastatin 20 mg
  Other Names: Lipitor
  Arms: Group A: Atorvastatin 20 mg
Drug: Placebo — Oral administration of placebo
  Arms: Group B: Placebo to Match (PTM)

SUMMARY:
Prospective randomized, multi-center, double blind placebo-controlled trial to assess the chemopreventive impact of atorvastatin (20 mg oral) vs placebo in up to 60 adults with advanced fibrosis at high risk of developing HCC.

DETAILED DESCRIPTION:
The study objective is to investigate the chemopreventive efficacy of atorvastatin (20 mg) on HCC risk compared to placebo in adults with advanced fibrosis (i.e. METAVIR fibrosis stage 3-4) and high-risk PLSec (defined by pre-randomization blood-based assay). HCC risk will be measured by changes in prognostic liver secretome signature (PLSec) risk score after oral administration of atorvastatin for 1 year with up to 5 years post-treatment of chart monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent
2. Male or female age > 18 years at time of consent
3. Clinically or histologically diagnosed advanced liver fibrosis or cirrhosis, as defined by one or more of the following:

   * Liver biopsy demonstrating advanced fibrosis or cirrhosis (METAVIR 3-4)
   * Fibroscan or MR elastography consistent with advanced fibrosis or cirrhosis
   * Imaging showing cirrhotic-appearing liver with signs of portal hypertension
   * Advanced fibrosis or cirrhosis documented clinically by a treating physician
4. High-risk for HCC at screening according to the FIB-4 index
5. PLSec score ≥ 3 measured in screening blood samples from the FIB-4-high individuals.
6. Liver imaging within 6 months of Day 1 is required in cirrhotic subjects only, to exclude HCC
7. Female subjects of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception
8. Willing and able to undergo protocol blood sampling
9. Subject must be able to comply with dosing instructions for study drug administration and able to complete study schedule of assessments

Exclusion Criteria:

1. Diagnosis of any of the following forms of chronic liver disease:

   * alpha-1-antitrypsin (A1AT) deficiency, Wilson disease, hemochromatosis, iron overload, prior known or suspected drug-induced liver injury (DILI)
   * Patients with PBC, PSC, AIH, or stable hemochromatosis may be included if their liver disease etiology overlaps with that of steatotic liver disease (SLD)
2. Current or prior history of any of the following:

   - Clinically significant illness or any other major medical disorder that in the opinion of the investigator, may interfere with subject treatment, assessment or compliance with the protocol
3. Known positivity for HIV infection
4. Active, untreated HCV infection

   - Patients with prior history of HCV who achieved sustained virologic response (SVR) >12 from Day 1 may be included in the study
5. Uncontrolled chronic HBV

   - Patients with well controlled disease with >12 months of stable medication use (or no medication use, in those persons for whom anti-HBV therapy is not indicated)
6. Clinical hepatic decompensation, defined as Child's Pugh class >B7 or C cirrhosis

   - Patients with Child's Pugh score of 7, class B, may be included in the study
7. History of biliary diversion
8. Solid organ transplant
9. Malignancy within the 5 years prior to screening, with the exception of specific cancers that have been cured by surgical resection (basal cell skin cancer, etc). Subjects under evaluation for possible malignancy are not eligible
10. Pregnant or Nursing Females (a negative serum pregnancy test is required at screening for WOCBP)
11. Life threatening SAE during the screening period
12. Subjects having the following laboratory parameters at screening

    * ALT > 10 x ULN
    * AST > 10 x ULN
    * Hemoglobin < 8.5 g/dl
    * Serum creatinine > 2.0 mg/dL
    * CK > 3x ULN
13. Females who may wish to become pregnant and/or plan to undergo egg harvesting during the study and up to 30 days of the last dose of study drug
14. WOCBP must abstain from breastfeeding and be willing to use effective birth control during through the week 4 post treatment follow-up visit
15. Clinically relevant alcohol or drug abuse within 12 months of screening
16. Use of any prohibited concomitant medications as described in Section 9.1.1
17. Use of a statin medication within 90 days of Day 1 visit

    - Subjects who are on a current statin at time of consent must be willing to undergo a 90-day washout period prior to randomization
18. Known hypersensitivity to atorvastatin
19. Current or planned participation in an investigational new drug (IND) trial from 30-days prior to randomization through the week 4 post treatment follow-up visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
Reduced magnitude of high-risk PLSec after treatment vs before treatment | 48 weeks
  The primary objective (primary endpoint) of this study is to determine the effect of atorvastatin compared with placebo on HCC risk level measured by change in serum-based prognostic liver secretome signature (PLSec) score (delta-PLSec).
  High-risk for HCC is indicated by a PLSec score of 3 or greater. Low-risk for HCC is indicated by a PLSec score below 3.

SECONDARY OUTCOMES:
Complete adverse event profile | 48 weeks
  Minimized toxicity in response to treatment based on NCI Common Terminology Criteria for Adverse Events (CTCAE) v.5 at least every 4 weeks to week 12 and at weeks 24, 36, and 48.
Complete profile of change in quality of life for patients | 48 weeks
  The investigators will assess the subjects' quality of life while on treatment using the Chronic Liver Disease Questionnaire (CLDQ). A Likert scale response format will be used for all items (n=29), and the overall CLDQ score will be obtained by adding scores for each item and dividing by the total number of items (n=29). The score ranges from 1 (most impairment) to 7 (least impairment).

OTHER OUTCOMES:
Exploratory Endpoint: Modulation of high-risk Prognostic Liver Signature (PLS) after treatment vs before treatment | 48 weeks
  The investigators will assess the significant magnitude of modulation in PLS-based HCC risk level calculated as the Combined Enrichment Score (CES) jointly measuring suppression of high-risk-associated genes and induction of low-risk-associated genes in the PLS.
  A negative CES indicates reduction of HCC risk level. The Mean CES between the treatment arms will be compared by using a two-sample t-test.
Exploratory Endpoint: Assessment of Pharmacokinetic (PK) Biomarkers of Atorvastatin | 48 weeks
  The investigators will assess the PK biomarkers of atorvastatin in serum from baseline and week 48. Serum atorvastatin concentration (ng/mL) will be measured between the atorvastatin group and placebo group.
Exploratory Endpoint: Assessment of Pharmacodynamic (PD) Biomarkers of Atorvastatin | 48 weeks
  The investigators will assess the PD biomarkers of atorvastatin in serum from baseline and week 48. Serum Low-Density Lipoprotein, or LDL (mg/mL) and total cholesterol concentration (mg/mL) will be measured between the atorvastatin group and placebo group.
Exploratory Endpoint: Assess the difference in HCC incidence rate between treatment groups | 288 weeks
  After subjects complete their on-treatment period, the study team will conduct a 5-year post-treatment observational study to examine the incidence rate of HCC between the atorvastatin group and the placebo group.
Exploratory Endpoint: Assessment of Immunohistochemical Markers of Pre/Neoplastic Foci | 48 weeks
  The investigators will assess the immunohistochemical markers of pre/neoplastic foci in formalin-fixed pre-treatment paraffin-embedded (FFPE) liver biopsy tissues. The investigators will measure the intensity of TAP cytoplasmic and nuclear staining by NIH ImageJ Software.
Exploratory Endpoint: Assessment of change in the proportion of high-risk patients defined by Prognostic Liver Secretome Signature (PLSec) score | 48 weeks
  In addition to the delta-PLSec assessed in the primary outcome, the investigators will assess the change in the proportion of subjects with high-risk PLSec (≥ 3) to low-risk PLSec (< 3) following treatment to be compared between the atorvastatin and placebo arms.
  The range of the PLSec score is 0 to 8. A higher PLSec score indicates a higher risk for hepatocellular carcinoma (HCC).

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Chung, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Dr. Raymond T. Chung. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: 1/2025-1/2026
Access Criteria: Researchers accessing IPD must be approved and have a data use agreement in place with Mass General Brigham to access the data.